CLINICAL TRIAL: NCT00822549
Title: Assessment of the Pharmacokinetic, Pharmacodynamic, Pharmacogenetic Relationships of Morphine and Metabolites After Severe Postoperative Pain in Adults
Brief Title: Pharmacokinetic, Pharmacodynamic and Pharmacogenetic of Morphine After Surgery
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOR 05038
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2009-01

CONDITIONS: Orthopaedic Surgery
Keywords: Morphine titration; Sub acute pain; Major orthopaedic surgery; Pharmacokinetics; Pharmacodynamics; Genetic polymorphism; PACU; Patients undergoing major scheduled orthopaedic surgery

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: all the patients included in the study received intravenous morphine in PACU and in the wards
  Interventions: Drug: intravenous morphine titration

INTERVENTIONS:
Drug: intravenous morphine titration — intravenous morphine titration

SUMMARY:
The main objective of this study is to improve our knowledge on the pharmacodynamic, pharmacokinetic, and pharmacogenetic relationships of morphine administered to relief severe postoperative pain. The analysis will encompass the efficacy (acute during titration and subacute during the first 24 hours) and adverse effects of morphine. Our purpose is also to better characterize the age- and sex-related differences which probably markedly differ between the two periods (acute vs sub acute).

DETAILED DESCRIPTION:
No previous study attempted to characterize the pharmacodynamic, pharmacokinetic, and pharmacogenetic relationships of morphine in the early postoperative period, whereas it is the main clinical situation for severe pain and a unique model for its study (not possible in the healthy volunteer). Indeed, intravenous titration of morphine is the first step for pain control in the postanesthesia care unit. Administration of intravenous boluses of morphine enables to obtain complete pain relief in 98% of the patients. We intend to study the effects of morphine (intravenous titration then patient-controlled intravenous administration (PCA) for 24 hours), perform dosages of plasma concentration of morphine an its main metabolites, and also study gene polymorphisms coding for main proteins involved in the pharmacokinetic and pharmacodynamic profile of morphine (hepatic metabolism, distribution and elimination, interaction with morphine receptor). Five hundred patients scheduled for major orthopedic surgery will be included in this prospective study. The main objective of this study is to improve our knowledge on the pharmacodynamic, pharmacokinetic, and pharmacogenetic relationships of morphine administered to relief severe postoperative pain. The analysis will encompass the efficacy (acute during titration and subacute during the first 24 hours) and adverse effects of morphine. Our purpose is also to better characterize the age- and sex-related differences which probably markedly differ between the two periods (acute vs subacute). We consider that this knowledge is important to confirm or not several important concepts currently used to define the appropriate analgesic regimen to control severe pain in the postoperative period.

ELIGIBILITY:
Inclusion criteria :

* scheduled major orthopedic surgery
* spine, hip or knee surgery
* Body weight between 50 and 100 kg
* Caucasians
* ASA status 1 to 3
* no cognitive dysfunction

Exclusion criteria :

* allergy or contraindication to morphine
* renal impairment (Cr Cl < 30 ml/min)
* severe hepatic impairment
* surgery performed under regional anaesthesia
* preoperative treatment including strong or weak opioids
* pregnancy, patients under 18 years, addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major orthopaedic surgery with severe postoperative pain. All the patients included in the study received intravenous morphine
Sampling Method: Non-Probability Sample
Enrollment: 438 (Actual)
Dates: Start 2006-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To improve our knowledge on the pharmacodynamic, pharmacokinetic and pharmacogenetic relationships of morphine administered after severe postoperative pain. | during the study

SECONDARY OUTCOMES:
- Relationships between morphine consumption, clinical events (efficacy or adverse effects) and morphine (and metabolites) blood concentrations. Immediate postoperative period (PACU) | Immediate postoperative period (PACU)
- Relationships between clinical events (pain relief, failure in pain relief, adverse effects) and genetic polymorphism. | Immediate postoperative period (PACU)
- Relationships between sub-acute clinical events and PK/PG profile. (on the wards at 24 hours after surgery) | on the wards at 24 hours after surgery
To better characterize the age- and sex-related differences which differ between acute and sub-acute periods. | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Aubrun, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital de la Pitié Salpêtrière, Paris, France

REFERENCES:
- [Derived] Aubrun F, Zahr N, Langeron O, Boccheciampe N, Cozic N, Belin L, Hulot JS, Khiami F, Riou B. Opioid-related genetic polymorphisms do not influence postoperative opioid requirement: A prospective observational study. Eur J Anaesthesiol. 2018 Jul;35(7):496-504. doi: 10.1097/EJA.0000000000000793. PMID 29474345